CLINICAL TRIAL: NCT04768712
Title: The Effect of Physical Activity on Physical Function, Falls and Bone Geometry - a Randomized Control Trial in Women With Manifest Osteoporosis
Brief Title: Effect of Physical Activity in Women With Manifest Osteporosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Mattias Lorentzon, Professor, Consultant, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VGFOUREG-81091
Record Dates: First submitted 2021-02-12; First posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weight bearing aerobic exercise (Experimental)
  Interventions: Behavioral: Weight bearing aerobic exercise
- Lifestyle counseling (No Intervention)

INTERVENTIONS:
Behavioral: Weight bearing aerobic exercise — Weight bearing aerobic exercise three times per week.
  Arms: Weight bearing aerobic exercise

SUMMARY:
Objectives: To investigate if a physical activity intervention (one year) can reduce the risk of falls (primary endpoint), improve physical function (balance and muscle strength) and cortical bone geometry as well as trabecular microarchitecture (secondary endpoints) in women, 70-80 years old, with manifest osteoporosis, treated with zoledronic acid, calcium and vitamin D.

Strategic goal: To include 200 patients (100 intervention and 100 controls) during 2010 and 2011 and randomize 100 patients to a one year physical activity intervention (3 hours weekly). The results will be published in an international scientific peer-review journal. All patients will receive standard medical treatment with calcium, vitamin D and yearly zoledronic acid.

Study rationale: The role of physical activity intervention has not previously been evaluated in patients with manifest osteoporosis and zoledronic acid treatment.

Methodology: Randomized controlled trial. All included patients (women 70-80 years of age) will have manifest osteoporosis, be treatment naïve, and will be treated on clinical indication with yearly infusions of zoledronic acid (approved treatment, for this patient category, by the Swedish Medical Products Agency). Patients with secondary osteoporosis, with disabilities, and with high levels of exercise at the baseline visit will be excluded. Intention to treat analysis will be used. Physical activity intervention includes 3 hours of weight bearing aerobic exercise per week, using a standardized program. Patients in both groups will be contacted monthly and asked about their exercise habits. Frequency of falls, physical activity level will be ascertained using questionnaires. Balance and muscle strength will be assessed using standardized tests. Bone geometry at the tibia diaphysis will be determined using an XCT2000 pQCT device (Stratec, Germany) and trabecular microarchitecture at the tibia metaphysis will be determined using an XtremeCT device (Scanco Medical AG, Switzerland). These examinations will be performed on all patients prior to the intervention and after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 70-80 years of age
* manifest osteoporosis, BMD T-score ≤2.5 SD at the lumbar spine and/or hip
* female
* walk without walking aid

Exclusion Criteria:

* male
* high level of exercise, ≥2 times/week, at baseline
* secondary osteoporosis
* previous treatment with bisphosphonate or other osteoporosis induced medicine

Ages: 70 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06-10 (Estimated); Primary Completion 2012-06-10 (Estimated); Study Completion 2012-06-10 (Actual)

PRIMARY OUTCOMES:
Propensity to fall | Through study completion, an average of 1 year
  Frequency of falls during time of intervention.

SECONDARY OUTCOMES:
Physical function (Balance and muscle strength) | Prior to the intervention and after the completion (an average of 1 year) of the study
Trabecular microarchitecture | Prior to the intervention and after the completion (an average of 1 year) of the study
Cortical bone geometry | Prior to the intervention and after the completion (an average of 1 year) of the study